CLINICAL TRIAL: NCT06866444
Title: Duloxetine Metabolism and Fibromyalgia
Acronym: DILIGENT
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jake Steenblik, Assistant Professor (Clinical), University of Utah
Other Study IDs: IRB_00167537
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Fibromyalgia; Duloxetine
Keywords: Duloxetine; Duloxetine metabolism
MeSH Terms: conditions — Fibromyalgia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — 10 mL blood sample will be obtained for a plasma duloxetine concentration and genotyping of CYP2D6 and CYP1A2.
  Blood samples will be obtained four hours after the morning dose with patients being nil per os to minimize the effect of gastric contents on duloxetine bioavailability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients treated with duloxetine for fibromyalgia: Adults 18+
  Meeting diagnostic criteria for Fibromyalgia
  Patients taking Duloxetine 60 mg/day for at least 8 weeks
  Interventions: Drug: Observational

INTERVENTIONS:
Drug: Observational — In a cohort of patients treated with duloxetine for fibromyalgia, participants vitals signs (blood pressure, heart rate, oxygen saturation level, temperature) will be taken as well as height and weight. Participants will fill out a questionnaire regarding their fibromyalgia diagnosis and symptoms. Lastly, participants will complete two sets of blood samples. One blood sample will evaluate genetic variants for duloxetine metabolizing capacity. The other sample will be used to analyze the level of concentration of duloxetine.

SUMMARY:
People with fibromyalgia report generalized body pain ("pain all over"), increased sensitivity to painful stimulation, chronic tiredness or low energy, sleep problems, and other physical and functional problems. The exact cause of the disorder is poorly understood, and treatment can be difficult.

The degree to which duloxetine is helpful for people with fibromyalgia varies greatly. For some people, it is very helpful for managing fibromyalgia symptoms. For others, people may not notice any benefit. Yet for some, it is a little helpful and the effect is noticeable only when people forget to take the medicine.

The purpose of this study is to collect data to better understand the relationship among gene types that control those enzymes, blood concentrations of duloxetine, and how it helps the symptoms.

DETAILED DESCRIPTION:
Study Purpose: To study the variability of response in patients with fibromyalgia to treatment with duloxetine

Duloxetine is a common FDA-approved pharmacotherapy for fibromyalgia. However, there is significant treatment response variability. Prior work has explored the role of liver drug-metabolizing enzymes CYP2D6 and CYP1A2 in the biotransformation of duloxetine. The genes coding for these enzymes have many variants; some variants are rapid metabolizers, whereas others are slow metabolizers of duloxetine. The different variants may contribute to the wide range of treatment responses to duloxetine among fibromyalgia patients. Supporting duloxetine metabolism as a contributor to drug response variability, researchers have measured plasma duloxetine concentrations following recommended dosing regimens and found concentrations to have substantial variability.

A strong correlation between an ultra-rapid duloxetine metabolizer with a poor response to duloxetine will provide useful information when formulating a treatment plan. Patients with a poor response to duloxetine phenotype may be better served by another serotonin norepinephrine reuptake inhibitor such as milnacipran. Early identification of those who would benefit from duloxetine will help a personalized approach to treating fibromyalgia and optimize the cost-effectiveness of pharmacological interventions.

Drug interactions with duloxetine that influence drug effect: An important consideration in characterizing duloxetine metabolism is to account for drug interactions that may inhibit or induce CYP1A2 or CYP2D6.

The main objective of this proposal is to conduct a feasibility study/pilot study to serve as the basis for a larger study where we refine our study methodology. In a cohort of patients treated with duloxetine for fibromyalgia, this study will measure:

(i) Symptoms of fibromyalgia using a validated questionnaire.

(ii) Duloxetine plasma concentrations.

(iii) Genotype CYP2D6 and CYP1A2 and correlate their plasma concentrations and genotype (rapid, normal, or slow metabolizer) with fibromyalgia symptoms.

Hypotheses:

(i) Patients with rapid or slow metabolizing variants will have low and high duloxetine plasma concentrations respectively.

(ii) Patients with rapid metabolizing variants will have ineffective treatment with duloxetine and patients with slow metabolizing variants will have signs and symptoms of effective treatment or duloxetine toxicity.

(iii) Patients who consume inducers or inhibitors of CYP2D6 or CYP1A2 will have low and high duloxetine plasma concentrations, respectively. Patients who consume inducers of CYP2D6 or CYP1A2 will have ineffective treatment with duloxetine, and patients that consume inhibitors of CYP2D6 or CYP1A2 will have signs and symptoms of effective treatment or duloxetine toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+
* Meeting diagnostic criteria for Fibromyalgia
* Patients taking Duloxetine 60 mg/day for at least 8 weeks

Exclusion Criteria:

* Pregnant patients per verbal confirmation
* Patients that have a history of physician diagnosed kidney or liver disfunction or history of renal dialysis.
* Patients requiring an interpreter to communicate
* Patient's with progressive illnesses other than fibromyalgia that have a chronic pain and fatigue component (e.g., cancer patients receiving antineoplastic treatment, Parkinson's disease, Multiple Sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Pain Management Center (PMC) at the University of Utah who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Duloxetine concentrations across metabolizer phenotypes, 3 groups | Obtained four hours after morning duloxetine dose.
  Metabolizer phenotypes will be separated into 3 groups based on diplotypes. Ultrarapid metabolizer phenotypes will be measured by having an activity score of greater than 2.0. Normal/intermediate metabolizer phenotypes will be measured by having an activity score between 1.0 to 2.0. Slow metabolizer phenotypes will be measured by having an activity score between 0.75 to 0.
Measure inhibitors and inducers of CYP1A2 and CYP2D6 in blood sample | Obtained four hours after the morning duloxetine dose.
  Inhibitors and inducers of CYP1A2 and CYP2D6 are defined by the Drug Interaction Flockhart Table. A strong inhibitor will be measured by ≥ 5-fold increase in plasma AUC or more than 80% decrease in clearance. A moderate inhibitor will be measured by 2 to 5-fold increase in the plasma AUC or 50-80% decrease in clearance.

SECONDARY OUTCOMES:
Symptoms of fibromyalgia | From start of study visit to end (approximately 2 hours).
  Measured by the Revised Fibromyalgia Impact Questionaire (FIQR) and ACR 2016 criteria for fibromyalgia. The FIQR is scored on a scale of 0-100, with higher scores (100) indicating a greater impact of fibromyalgia (worst outcome) and lower scores (0) indicating a lesser impact of fibromyalgia (better outcome).
Vital signs, heart rate | One time at the start of the study visit.
  Heart rate (bpm) will be recorded.
Vital signs, noninvasive blood pressure | One time at the start of the study visit.
  Blood pressure (mmHg) readings will be recorded.
Vital signs, oxygen hemoglobin saturation | One time at the start of the study visit.
  Oxygen hemoglobin saturation (Sp02 using pulse oximeter) will be recorded.
Vital signs, temperature | One time at the start of the study visit.
  Temperature (Celcius) will be recorded.
Vital signs, respiratory rate | One time at the start of the study visit.
  Respiratory rate will be recorded (via observation for 1 minute).

CONTACTS AND LOCATIONS:
Overall Officials: Jake Steenblick, DNP, Principal Investigator — University of Utah
Locations (1):
- Pain Management Center and Pain Research Center at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No